CLINICAL TRIAL: NCT07043075
Title: First-in-Human (FIH) Study on the Feasibility and Safety of the TaviPilot Augmented Reality Guidance Software Operated in Parallel Setup During Transcatheter Aortic Valve Implantation (TAVI) Without Influencing Clinical Decision-Making
Brief Title: First-in-Human (FIH) Study on the Feasibility and Safety of the TaviPilot Augmented Reality Guidance Software
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caranx Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 55002-01
Record Dates: First submitted 2025-06-04; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAVR procedure with TAVIPILOT (investigational medical device) (Experimental)
  Interventions: Device: TAVR using a guidance software

INTERVENTIONS:
Device: TAVR using a guidance software — TAVR procedure with TAVIPILOT augmented reality guidance software operating in parallel on a separate screen in a blind setup, enabling clinicians to assess the analysis and recommendations provided by the software, either immediately after valve deployment or following the completion of the procedure.

SUMMARY:
The trial aims to evaluate the feasibility and safety of Caranx Medical TAVIPILOT augmented reality guidance software during Transcatheter Aortic Valve Replacement Procedures.

DETAILED DESCRIPTION:
The study is a prospective mono-center single-arm study to evaluate primarily the feasibility and safety of TAVIPILOT augmented reality guidance software during Transcatheter Aortic Valve Replacement Procedures (TAVR) for severe aortic stenosis. A series of parameters will be analysed to determine whether TAVIPILOT is a safe tool for valve positioning.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥65
2. Indicated for transfemoral TAVR for severe aortic stenosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Investigational Device Safety | Peroperative
  Exploratory evaluation of the technical robustness of the Investigational Device (TaviPilot Software) by evaluating the occurence of malfunctions while operating passively in parallel of the clinical procedure

SECONDARY OUTCOMES:
Investigational Device Performance | Peroperative
  Assess the performance of the device by comparing the valve implantation depth measured by the TaviPilot Software with the depth estimated by the investigator who performed the procedure.
Investigational Device Performance | Peroperative
  Assessment of clinician satisfaction related to device usability and performance using custom made questionnaires

IPD SHARING:
Plan to Share IPD: No